CLINICAL TRIAL: NCT03547791
Title: Effects of Antenatal Corticosteroid in Twin Neonates With Late Preterm Birth: Study Protocol for a Randomized Controlled Trial
Brief Title: Effects of ACS in Twin With LPB: Study Protocol for a RCT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Twin_RCT_2018
Record Dates: First submitted 2018-03-29; First posted 2018-06-06 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Twin Pregnancy, Antepartum Condition or Complication
Keywords: Antenatal corticosteroid; Twin pregnancies; Respiratory morbidity; Randomized controlled trial
MeSH Terms: interventions — betamethasone sodium phosphate; Saline Solution

STUDY DESIGN:
Intervention Model Description: In this multi-center, double-blind, randomized, placebo-controlled trial, women who are at risk for late preterm birth (34+0wks-36+5wks) will be enrolled and randomly assigned to two groups receiving betamethasone(ACS) or placebo.
Who Masked: Participant, Care Provider
Masking Description: Enrolled women will be randomly assigned in a 1:1 ratio to ACS (Group 1) or placebo (Group 2). The randomization will be done by web-based randomization system which is operated by medical research collaborating center of Seoul National University Hospital. The ACS or placebo will be prepared by unblended researchers [clinical trial pharmacy]. Unblinded researchers will be designated at the beginning of this trial, and they will not participate in the subsequent process of data management and data analysis. Neither the enrolled pregnant women nor the other investigators (except predeterminate unblinded researchers) will be aware of the result of random assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACS (Group 1) (Active Comparator): Intramuscular injection of betamethason sodium phosphate 12mg (3ml) twice 24hours apart
  Interventions: Drug: Betamethason Sodium Phosphate
- Placebo (Group 2) (Placebo Comparator): Intramuscular injection of normal saline 3ml twice 24hours apart
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Betamethason Sodium Phosphate — The antecorticosteroid that will be administered to Group 1 is betamethasone, produced by Dawon Parm(Korea). It contains betamethason sodium phosphate 5.2mg(Betamethasone 4.0mg) in 1 ample(1mL). Each drug is carried in a syringe by pharmacist who does not participate in study after the patient was enrolled in the study and administered to the patient twice 24hours apart.
  Other Names: ACS
  Arms: ACS (Group 1)
Drug: Normal saline — Intramuscular injection of normal saline 3ml twice 24hours apart
  Other Names: NS
  Arms: Placebo (Group 2)

SUMMARY:
This study will be the first study that evaluates the effectiveness of antenatal corticosteroid (ACS) in late preterm twin neonates.

DETAILED DESCRIPTION:
Antenatal corticosteroid (ACS) has been proven to prevent adverse outcomes including respiratory morbidities in preterm neonates before 34 weeks of gestations. Recently, it has been suggested that ACS may be also effective for reduction of respiratory complications in singleton late preterm pregnancies. On the contrary, there is a paucity of information regarding the effectiveness of ACS in twin neonates with late preterm birth, and nowadays guidelines are recommending the use of ACS in twin pregnancies based on the evidences in singleton pregnancies. However, the effect of ACS in twin needs to be determined, because the rate of neonatal morbidities in twin preterm neonates seems to be different from that in singleton neonates. This study aims to determine the effectiveness of ACS in late preterm twin neonates.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age over 18 years
* (2) Twin pregnant women at 34weeks 0days to 36weeks 5days of gestation
* (3) At risk for preterm birth such as preterm labor, preterm prematrue rupture of membrane or maternal-fetal indications that need preterm delivery. Preterm labor is defined as regular uterine contractions with or without the following symptoms; pelvic pressure, backache, increased vaginal discharge, menstrual-like cramps, bleeding/show, cervical changes
* (4) Availability of written informed consent.

Exclusion Criteria:

* (1) Gestational age before 34weeks 0days or after 36weeks 6days
* (2) Lethal major fetal anomaly, fetal distress or fetal death in utero
* (3) Expected to deliver within 12 hours; for example, advanced cervical dilatation (>8cm) in preterm labor or active phase labor (cervical dilatation>4cm) in preterm premature rupture of membranes
* (4) History of a previous administration of ACS before 34weeks of gestation for fetal lung maturation
* (5) Administration of systemic steroid for medical indications
* (6)Diagnosis of clinical chorioamnionitis Fever >37.8 and the presence of two more following conditions: uterine tenderness, foul-odored vaginal discharge, maternal leukocytosis(>1500), maternal tachycardia(>100) or fetal tachycardia(>160)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 848 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory morbidity | 72 hours after birth
  NICU admission, Continuous positive airway pressure, High flow nasal cannula for ≥12 continuous hours, Fraction of inspired oxygen of ≥ 0.3, Mechanical ventilation use, ECMO use and Stillbirth or neonatal death within 72hours after death

SECONDARY OUTCOMES:
Maternal complication | 72 hours after birth
  Chorioamnionitis and Postpartum endometritis
Respiratory distress syndrome | 72 hours after birth
  Presence of clinical signs of respiratory distress (tachypnea, retractions, flaring, grunting, or cyanosis), with a requirement for supplemental oxygen with a fraction of inspired oxygen of more than 0.21 and a chest radiograph showing hypoaeration and reticulogranular infiltrates
Transient tachypnea of the newborn, apnea | 72 hours after birth
  Tachypnea occurred in the absence of chest radiography or with a radiograph that was normal or showed signs of increased perihilar interstitial markings and resolved within 72 hours
Need for resuscitation at birth | at birth
  any intervention in the first 30 minutes other than blow-by oxygen
Surfactant use | 28 days after birth
  Surfactant use
Bronchopulmonary dysplasia;BPD | 28 days after birth
  Requirement for supplemental oxygen with a fraction of inspired oxygen of more than 0.21 for the first 28 days of life

OTHER OUTCOMES:
Necrotizing enterocolitis (NEC) | 28 days after birth
  meconium plug syndrome or confirmed NEC by pathohistology or operation finding
Birth weight | at birth
  neonatal body weight
1 minute, 5minute Apgar score | at birth
  evaluation(scoring) of neonatal appearance, pulse, grimace, activity, respiration 1 minute and 5minute after birth
Hypoglycemia | 28 days after birth
  Glucose < 40 mg%
Hyperbilirubinemia | 28 days after birth
  Peak total bilirubin of at least 15 mg% or the use of phototherapy
Feeding difficulty | 28 days after birth
  Inability to take all feeds (po), i.e. requiring gavage feeds or IV supplementation. In addition, time to first feed (po) will be recorded
Neonatal infectious morbidity | 28 days after birth
  Sepsis, Suspected sepsis and Pneumonia
Seizures / encephalopathy | 28 days after birth
  Witnessed seizure
Hospital day of NICU admission | 28 days after birth
  Includes need for NICU or intermediate care admission and length of stay if admitted

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee SM, Park HS, Choi SR, Lee J, Kim HJ, Park JY, Oh KJ, Cho GJ, Oh MJ, Chung JH, Kim SM, Kim BJ, Kim SY, Hong S, Jung YM, Lee SJ, Seong JS, Kim H, Oh S, Lee J, Jin YR, Kim JH, Cho HY, Park CW, Park JS, Jun JK. Antenatal Corticosteroid in Twin-Pregnant Women at Risk of Late Preterm Delivery: A Randomized Clinical Trial. JAMA Pediatr. 2025 Dec 1;179(12):1275-1282. doi: 10.1001/jamapediatrics.2025.3284. PMID 40982289
- [Derived] McGoldrick E, Stewart F, Parker R, Dalziel SR. Antenatal corticosteroids for accelerating fetal lung maturation for women at risk of preterm birth. Cochrane Database Syst Rev. 2020 Dec 25;12(12):CD004454. doi: 10.1002/14651858.CD004454.pub4. PMID 33368142
- [Derived] Hong S, Lee SM, Kwak DW, Lee J, Kim SY, Oh JW, Oh S, Park CW, Park JS, Chung JH, Jun JK. Effects of antenatal corticosteroids in twin neonates with late preterm birth (ACTWIN [Antenatal Corticosteroids in TWIN late preterm neonates] trial): study protocol for a randomized controlled trial. BMC Pregnancy Childbirth. 2019 Apr 3;19(1):114. doi: 10.1186/s12884-019-2235-5. PMID 30943910